CLINICAL TRIAL: NCT05563272
Title: Phase 2, Multicenter, Open-Label Study of 89Zr-girentuximab for PET/CT Imaging of Tumors Likely to Express High Levels of CAIX
Brief Title: 89Zr-girentuximab for PET Imaging of CAIX Positive Solid Tumors
Acronym: STARBURST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Indication scouting for TLX250-CDx will continue in theranostic studies, with a therapeutic component in the study design.
Sponsor: Telix Pharmaceuticals (Innovations) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 89Zr-TLX250-005
Record Dates: First submitted 2022-09-23; First posted 2022-10-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Glioblastoma Multiforme; Cholangiocarcinoma; Hepatocellular Carcinoma; Head and Neck Squamous Cell Carcinoma; Nasopharyngeal Carcinoma; Non Small Cell Lung Cancer; Small Cell Lung Cancer; Epithelial Ovarian Cancer; Pancreatic Ductal Adenocarcinoma; Soft Tissue Sarcoma; Gastric Adenocarcinoma; Malignant Mesothelioma (MM); Von Hippel Lindau; Bladder Cancer; Bladder Urothelial Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Glioblastoma; Cholangiocarcinoma; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial; Sarcoma; Mesothelioma, Malignant; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-TLX250 (Experimental)
  Interventions: Diagnostic Test: 89Zr-girentuximab for PET/CT imaging of CAIX positive tumors

INTERVENTIONS:
Diagnostic Test: 89Zr-girentuximab for PET/CT imaging of CAIX positive tumors — On Day 0, participants will receive a single administration of 89Zr-girentuximab (37 Megabecquerel (MBq) [1mCi] ± 10%, containing a mass dose of 10 mg of girentuximab).

SUMMARY:
A prospective, open-label, phase 2 study to explore CAIX expression through 89Zirconium-labelled girentuximab deferoxamine (89Zr-girentuximab) PET/CT imaging in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the following criteria:

1. Written and voluntarily given Informed Consent.
2. Male or female ≥18 years of age at time of consent.
3. Have the capacity to understand the study and be willing and able to comply with all protocol requirements.
4. Participants must have proven tumors of the following types, but not limited to:

   * Cervical cancer;
   * Colorectal cancer;
   * Esophageal SCC and esophageal/esophagogastric junction adenocarcinoma;
   * Gastric adenocarcinoma;
   * GBM;
   * Head and neck SCC and nasopharyngeal carcinoma;
   * cholangiocarcinoma and hepatocellular carcinoma;
   * non-small cell lung cancer;
   * small cell lung cancer;
   * epithelial ovarian carcinoma;
   * pancreatic ductal adenocarcinoma;
   * Soft tissue sarcoma;
   * malignant mesothelioma;
   * confirmed diagnosis of VHL disease with VHL germline alteration and at least one VHL-related lesion.
5. Have at least one non-central nervous system (CNS), measurable target lesion as defined per RECIST 1.1 and documented by SOC conventional imaging, performed within 60 days (+14 days) prior to Day 0 (excepting participants with GBM or hemangioblastoma, given that all lesions may be in the CNS, such lesions assessed by RANO);
6. Have agreed not to receive another investigational product while participating in the present study, defined as signing the informed consent form (ICF), until completion of the last study visit;
7. Have negative serum pregnancy tests if a female of childbearing potential at screening and have a confirmatory negative urine pregnancy test result within 24 hours prior to receiving investigational product. Female participants of non-child- bearing potential must provide evidence by fulfilling one of the following criteria at screening:

   * Be post-menopausal, defined as more than 50 years of age and amenorrheic for at least 12 months since cessation of all exogenous hormonal treatments;
   * Be a woman under 50 years of age and considered postmenopausal given amenorrhea for 12 months or more since cessation of exogenous hormonal treatments and having luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range by institutional SOC;
   * Have documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation; and
8. Have consented to practice highly effective method of contraception until a minimum of 42 days after 89Zr-girentuximab administration

Exclusion Criteria

Participants will be excluded from participation in the study if one or more of the following criteria are met:

1. Have been administered any radionuclide within 10 half-lives (of the radionuclide) prior to the intended administration of 89Zr-girentuximab (i.e., within 10 half-lives of Day 0);
2. Have been exposed to any CAIX targeting compound (diagnostic/therapeutic) in the prior 3 months;
3. Have any serious non-malignant disease (e.g., psychiatric, infectious, autoimmune or metabolic) that may interfere with the objectives of the study or with the safety or compliance of the participant, as judged by the Investigator;
4. Have any clinically significant abnormalities detected during screening laboratory tests or physical exam that, in the opinion of the Investigator, would adversely affect the participant's ability to participate in the study;
5. Have a mental impairment that may compromise the ability to give Informed Consent and comply with the requirements of the study;
6. Have been exposed to any antineoplastic treatment from Day 0 (89Zr-girentuximab dosing) to completion of 89Zr-girentuximab PET/CT imaging (Day 5 ± 2 days);
7. Be a female who is pregnant or breastfeeding;
8. Have a known allergy, hypersensitivity, or intolerance to girentuximab, desferrioxamine (DFO), or any of the components of the investigational agent;
9. Have renal insufficiency with a glomerular filtration rate (GFR) ≤45 milliliters/min/1.73m2
10. Be a vulnerable participant (e.g., being in detention).

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of 89Zr-girentuximab uptake within individual tumor deposits | Single diagnostic administration, followed by a diagnostic scan on Day 5 ± 2 days. This assessment will be conducted throughout the patient dosing and imaging period, an average of 18 months
  This outcome will be evaluated on all patients by using a PET/CT machine to qualitatively assess (yes / no) the uptake of the 89Zr-girentuximab uptake within individual tumor deposits.
Quantitative assessment of 89Zr-girentuximab uptake within individual tumor deposits | Single diagnostic administration, followed by a diagnostic scan on Day 5 ± 2 days. This assessment will be conducted throughout the patient dosing and imaging period, an average of 18 months
  This outcome will be evaluated on all patients by using a PET/CT machine to quantitatively assess the uptake of the 89Zr-girentuximab uptake within individual tumor deposits.

SECONDARY OUTCOMES:
To evaluate safety parameter of Heart rate in patients administered with 89Zr-girentuximab | Patients will be evaluated for the period up to imaging following administration of 89Zr-girentuximab, at most 7 days.
  This outcome will be measured as beats per minute on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria
To evaluate safety parameter of blood pressure in patients administered with 89Zr-girentuximab. | Patients will be evaluated for the period up to imaging following administration of 89Zr-girentuximab, up to 7 days.
  This outcome will be measured as mmHg on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria
To evaluate safety parameter related to Liver function in patients administered 89Zr-girentuximab | Patients will be evaluated for the period up to imaging following administration of 89Zr-girentuximab, up to 7 days.
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.
To evaluate safety parameter related to Renal function in patients administered 89Zr-girentuximab | Patients will be evaluated for the period up to imaging following administration of 89Zr-girentuximab, up to 7 days.
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.
To evaluate safety parameter related to Full Blood Count in patients administered 89Zr-girentuximab | Patients will be evaluated for the period up to imaging following administration of 89Zr-girentuximab, up to 7 days.
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, Los Angeles(UCLA), Los Angeles, California
  - Biogenix Molecular, LLC, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Munson Medical Center, Traverse City, Michigan
  - University Hospitals Cleveland Medical Center (UHCMC), Cleveland, Ohio
  - Kettering Health Research Institute, Kettering, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Austin Radiological Association (ARA), Austin, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Inland Imaging, Spokane, Washington